CLINICAL TRIAL: NCT02870582
Title: Efficacy and Safety of Donafenib in Patients With Previously Treated Metastatic Colorectal Cancer:a Controlled,Multicentre,Randomised, Phase 3 Trial
Brief Title: Donafenib for Previously Treated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZGDC3
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — donafenib; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Donafenib (Experimental): Donafenib 300mg bid on 1-21 days of each 28 days cycle.
  Interventions: Drug: Donafenib
- Placebo (Placebo Comparator): Placebo 300mg bid on 1-21days of each 28 days cycle.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donafenib — treatment drug
  Other Names: CM4307
  Arms: Donafenib
Drug: Placebo — Best support treatment
  Other Names: Controlled
  Arms: Placebo

SUMMARY:
The investigators do the clinical trial (patients with metastatic colorectal cancer treated with donafenib/placebo after failure of standard therapy) to assess efficacy and safety of donafenib in patients with metastatic colorectal cancer, progressing after all approved standard therapies.

DETAILED DESCRIPTION:
The study is a randomization,multicentre, phase 3 study recruiting 510 patients. Patients were eligible to participate when they have histological or cytological documentation of adenocarcinoma of the colon or rectum. They must have received locally and currently approved standard therapies and to have disease progression during or within 3 months after the last administration of the last standard therapy or to have stopped standard therapy because of unacceptable toxic effects. The available standard therapies have to include as many of the following as were licensed: a fluoropyrimidine,oxaliplatin,irinotecan.

All patients receive best supportive care, excluding other investigational antitumour agents or antineoplastic chemotherapy, hormonal therapy, or immunotherapy.

Patients receive oral donafenib 300mg (CM4307) on days 1-21 of each 4 weeks cycle until disease progression,death,or the unacceptable toxic effects.The primary endpoint is overall survival.The second endpoint is progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of adenocarcinoma of the colon or rectum;
* Subjects with metastatic colorectal cancer and must have progressed during or within 3 months following the last administration of approved standard therapies which must include a fluoropyrimidine, oxaliplatin and irinotecan:

  1. Subjects treated with oxaliplatin in an adjuvant setting should have progressed during or within 6 months of completion of adjuvant therapy;
  2. Subjects who progress more than 6 months after completion of oxaliplatin containing adjuvant treatment must be retreated with oxaliplatin-based therapy to be eligible;
  3. Subjects who have withdrawn from standard treatment due to unacceptable toxicity warranting discontinuation of treatment and precluding retreatment with the same agent prior to progression of disease will also be allowed into the study;
  4. Subjects may have received prior treatment with bevacizumab and/or cetuximab/panitumumab.
* Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to randomization EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 1;
* Life expectancy of at least 3 months;
* Adequate bone marrow, liver and renal function as assessed by the laboratory required by protocol conducted within 7 days before randomization (platelets >80× 109/L, neutrophil > 1.5 × 109/L, Hb≥85g/L, serum creatinine ≤ 1.5×ULN, total bilirubin ≤ 1.5×ULN, and serum transaminase≤2.5×ULN or ≤5.0ULN if liver involvement);

Exclusion Criteria:

* Prior treatment with TKIs.
* Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to randomization EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* Subjects who have no evaluable lesion except Pleural effusion, ascites or bone metastases lesion;
* Major surgery have been completed within 4 weeks before the first dose of study medicine.
* Subjects who have open wounds, active ulcers or plural stomata;
* Subjects who have completed radiotherapy or systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and hormonal therapy during this trial or within 4 weeks before the first dose of study medicine;
* Cardiological disease including Congestive heart failure, Unstable angina, Myocardial infarction, Cardiac arrhythmias requiring anti-arrhythmic therapy.
* Pleural effusion or ascites that causes respiratory compromise.
* Arterial or venous thrombotic or embolic events.
* Any history of or currently known brain metastases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From randomization of the first subject until 316 death events observed, up to 2 years
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | From randomization of the first subject until 316 death events observed, up to 2 years
  PFS was defined as the time from date of randomization to disease progression radiological or death due to any cause, whichever occurs first. Subjects without progression or death at the time of analysis were censored at their last date of tumor evaluation.
Disease Control Rate (DCR) | From randomization of the first subject until 316 death events observed, up to 2 years
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD); CR, PR, or SD had to be maintained for at least 28 days from the first demonstration of that rating)
Safety variables will be summarized using descriptive statistics based on adverse events collection | From randomization of the first subject until 316 death events observed, up to 2 years
  AE evaluated by CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Bi Feng, MD, Study Chair — West China Hospital; Xu Jianming, MD, Study Chair — The Affiliated Hospital of Military Medical Sciences
Locations (2):
- China (2):
  - the 307th Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - West China Hospital Sichuan, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No
No plan to share date of the trial